CLINICAL TRIAL: NCT00487409
Title: A Randomized Trial Comparing Outcomes for the LigaSure and Disposable Stapling Instruments for Laparoscopic Surgery
Brief Title: Random Comparison of LigaSure and Disposable Staples for Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Principal Investigator, Conor Delaney, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-06-33
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Colonic Diseases; Rectal Diseases
Keywords: Ulcerative colitis; Crohn's disease; Colorectal polyps; Colorectal malignancy; Endometriosis; Diverticulitis; Colonic inertia
MeSH Terms: conditions — Colonic Diseases; Rectal Diseases; Colitis, Ulcerative; Crohn Disease; Endometriosis; Diverticulitis; Constipation | interventions — Sutures; Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Standard of Care
  Interventions: Procedure: Disposable stapling instruments
- Group B (Other): Standard of Care
  Interventions: Procedure: Bipolar electrosurgical generator and instruments

INTERVENTIONS:
Procedure: Bipolar electrosurgical generator and instruments — laparoscopic colectomy using the Ligasure device
  Other Names: Ligasure Device
  Arms: Group B
Procedure: Disposable stapling instruments — laparoscopic colectomy using clips, cautery and stapler
  Other Names: Staples or Clips
  Arms: Group A

SUMMARY:
The purpose of this research is to compare two different standard of care surgical methods for the following large bowel (colon) procedures: laparoscopic right colectomy, total colectomy, and left colectomy. The study will compare electrocautery, used with surgical clips and/or surgical staplers, and the Ligasure vessel sealer. The investigators will be looking at which procedure is faster and more cost efficient and the investigators will calculate hospital expenses for the two groups to make comparisons.

DETAILED DESCRIPTION:
The application of laparoscopic surgery has expanded over the last decade to include many complex abdominal procedures that have traditionally been performed through a laparotomic incision. The widespread acceptance and utilization of laparoscopy has directly resulted in a continuing need to develop both new techniques and ancillary surgical instrumentation.

Laparoscopic instruments that provide adequate hemostasis and allow for precise dissection of tissues are needed for a safe and efficient operation. Furthermore, as new devices emerge and the volume of laparoscopic cases increases the importance of cost and ergonomically sound instrumentation have become apparent.

The safety and efficacy of laparoscopic colectomy for benign disease has been demonstrated by several case series over the last decade. The advantages of smaller wounds, shorter ileus, earlier resumption of dietary intake, and reductions in hospital stay have been consistently reported as the major benefits of this approach. More recently, in a multi-center randomized prospective trial laparoscopic colectomy for curable cancer resulted in equivalent cancer related survival to open colectomy when performed by experienced surgeons. Adherence to standard cancer resection techniques including but not limited to complete exploration of the abdomen, adequate proximal and distal margins, ligation of the major vessels at their respective origins, containment and careful tissue handling, and en bloc resection with negative tumor margins using the laparoscopic approach resulted in acceptable outcomes.

The advantages of standardized surgical technique's for laparoscopic colectomy that were discussed in this multicenter trial were well outlined in one previous study. This study retrospectively reviewed a consecutive series of patients undergoing laparoscopic sigmoid colectomy from 1999 to 2001 at a single institution. The potential benefits of a standardized technique included 1) standardization of surgical instrument sets, 2) definition of benchmarks for the decision to convert before inappropriate investments in time and equipment, and 3) provision of an easily transferred skill set for residents in training.

Despite the obvious value of this standardized approach, a variety of techniques and laparoscopic instruments for tissue dissection and coagulation are currently utilized. These options include laparoscopic staplers, lap clip appliers, suture ligature, electrothermal bipolar vessel sealers, electric cautery, and ultrasonic shears. Dissection, coagulation, and the division of the mesocolon and mesorectum during laparoscopy, continue to represent a technical and hemostatic challenge. When dealing with inflamed tissues, as in diverticulitis or inflammatory bowel disease, or when the mesocolon and mesorectum are fatty, reliable hemostasis is not always easy to obtain. Concerning tissue dissection and coagulation, electrosurgery, widely implemented in open surgery, has displayed some complications and limits related to minimally invasive techniques. The search for safer multidimensional instruments has led to the development of both the ultrasonic dissector(UCS), (Harmonic Scalpel, Ultracision, Ethicon Endosurgery Inc., Cincinnati, OH) and the endoscopic Ligasure (LIG or EBVS), (Valleylab, Boulder, CO).

Use of ultrasonic dissection in colorectal laparoscopic surgery has recently been reviewed retrospectively in two studies. Both studies concluded that ultrasonic dissection was safe and effective. A prospective randomized clinical trial also demonstrated that use of UCS provided the advantage of a decreased blood loss when compared with ES without and any increase in morbidity.

Recently an electrothermal bipolar vessel sealer, (EBVS) (Ligasure, Valleylab, Boulder, CO, USA) was developed for both laparoscopic and open procedures as an alternative to suture ligatures, hemoclips, staplers and ultrasonic coagulator's for ligating vessels, and tissue bundles. The EBVS is approved by the Food and Drug Administration to seal vessels up to 7mm in diameter. It does so by applying high current and low voltage, which differs from the energy used in standard monopolar and bipolar cautery. This unique form of energy denatures collagen and elastin within the vessel wall and surrounding connective tissue. The addition of extreme pressure applied by the instrument, which also differs from other energy sources, causes the denatured protein to reform, with the vessel walls in apposition. Clinically, the result is a nearly translucent "seal" that may be transected. The Ligasure device has been used in all types of gastrointestinal surgery including small and large bowel resection, gastrectomy, pancreatectomy, splenectomy, esophagogastric devascularization for portal hypertension, and transplantation. To date, the device appears to be cost effective in teaching institutions when used in difficult open and laparoscopic surgery.

The initial results with the EBVS and colorectal surgery were from a prospective review of 98 cases by a single surgeon from 1998 to 2000. These included both laparoscopic and open cases and involved 53 colon resections. No postoperative hemorrhagic complication occurred and there was an estimated mean reduction in operative time of 39 minutes. Additionally, the same authors' applied the ligasure technology to a pig animal model and consistently reported no evidence of postoperative bleeding. They concluded that the EBVS was safe and effective and may potentially reduce operative times.

A second study, also a retrospective analysis, compared Ligasure to an ultrasonic coagulator for total abdominal colectomy in 15 patients with ulcerative colitis. The procedure using Ligasure reduced the operating time, intraoperative bleeding and operator's stress in comparison with ultrasonic coagulation.

A third study, another retrospective comparative model, was conducted to address the differences between EBVS and ultrasonic shears for laparoscopic transverse and sigmoid colectomy. The study included 30 patients and found that the incidence of rebleeding was significantly lower in the EBVS group than in the the UCS group for both surgical procedures. In addition the required time for mesocolon dissection was also significantly shorter when the EBVS was used.

The only prospective randomized study with Ligasure and laparoscopic colorectal surgery addressed the speed, reliability and cost to guide surgeons in their choice for intracorporeal pedicle ligation. This study involved both straight laparoscopy and hand-assisted laparoscopy and compared laparoscopic vascular staplers and disposable clip appliers with the Ligasure Atlas during elective right, left, and total colectomy. Cases were stratified by procedure and failure was defined as any bleeding after pedicle ligation. 100 patients were included in the study and the Ligasure atlas was found to be more cost effective and associated with lower failure rates.

Significance and Purpose The utilization and safety of surgical staplers and disposable clips for laparoscopic colectomy is established and has been adopted by the majority of surgeon's performing these procedures. Although the growing evidence supporting the application of Ligasure to laparoscopic colorectal surgery has demonstrated its safety and efficiency, most of the studies have been limited by sample size and their retrospective nature. There also have been several questions left unanswered. A standardized approach for laparoscopic right, total, and left colectomy has never been substantiated by any prospective study. Furthermore, the difficult and somewhat dangerous steps involved with division of the mesorectum during both laparoscopic sigmoid colectomy and low anterior resection have not been appropriately evaluated.

The objective of this study is to determine the best technical approach to laparoscopic right, total, and left colectomy by comparing the utilization of the Ligasure device to electrocautery with the application of surgical clips and/or surgical stapler's. To answer this question the investigators will compare each approach regarding tissue dissection, colonic mobilization and pedicle ligation. Safety, cost, operative time, time to pedicle ligation and hemostasis will be objectively measured in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have benign or malignant colonic or rectal disease that mandate resection and are approached laparoscopically. Potential indications or conditions include ulcerative colitis, Crohn's disease, colorectal polyps, colorectal malignancy, endometriosis, diverticulitis, and colonic inertia
* Subjects who are 18 years of age and older
* Subjects of either sex
* Subjects who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent

Exclusion Criteria:

* Subjects who undergo conversion to the open approach before mobilization of the colon or pedicle ligation will be excluded from the analysis
* Subjects who are pregnant
* Subjects who have undergone a previous colectomy
* Subjects with a medical condition that may interfere with the evaluation of safety or effectiveness of the study device
* Subjects who have another condition that in the opinion of the investigator precludes further participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
this study will evaluate the surgical approach using the Ligasure device at six weeks post operative. | 6 weeks post-op
  The objective of this study is to determine the best technical approach to laparoscopic right total and left colectomy by comparing the utilization of the Ligasure device to electrocautery with the application of surgical clips and or surgical staples. Safety, cost, operative time, time to pedicle ligation and hemostasis will be objectively measured in each treatment group.

SECONDARY OUTCOMES:
Will evaluate the surgical approach using electrocautery with surgical clips and staples | 6 weeks post op
  The objective of this study is to determine the best technical approach to laparoscopic right total and left colectomy by comparing the utilization of the Ligasure device to electrocautery with the application of surgical clips and or surgical staples. Safety, cost, operative time, time to pedicle ligation and hemostasis will be objectively measured in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Conor P. Delaney, MD, PhD, Principal Investigator — University Hospitals of Cleveland/ Institute for Surgical Innovation
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Adamina M, Champagne BJ, Hoffman L, Ermlich MB, Delaney CP. Randomized clinical trial comparing the cost and effectiveness of bipolar vessel sealers versus clips and vascular staplers for laparoscopic colorectal resection. Br J Surg. 2011 Dec;98(12):1703-12. doi: 10.1002/bjs.7679. Epub 2011 Oct 13. PMID 21997317